CLINICAL TRIAL: NCT05452876
Title: Alberta Back Care Pathway (ABCp)
Acronym: ABCp
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Chiropractic Research Foundation (Unknown); Bone and Joint Health SCN (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00105576
Record Dates: First submitted 2022-05-09; First posted 2022-07-11 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: non-randomized, stepped-wedge, multi-clinic (cluster) prospective cohort design having multiple controls within a primary care setting
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABCp (Experimental): The patient sees MD that follows ABCp, patient then enrolls in ABCp intervention based on MD's categorization of low back pain.
  Interventions: Other: ABCp
- Usual Care (Active Comparator): The patient receives "usual care" at the clinical site.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: ABCp — Intervention is a care pathway that helps primary care physicians categorize back pain patients with each category having preferred interventions.
  Arms: ABCp
Other: Usual Care — Standard of care treatment
  Arms: Usual Care

SUMMARY:
Every year, the pain, disability, addiction, and expense associated with LBP increase in Alberta. This escalation is largely because most people with LBP seek care from family physicians who are unable to provide effective, guideline-based interventions due to three recognized barriers: 1) a lack of training, 2) a lack of no (or low) cost access to these interventions and 3) a lack of physician time and reimbursement to deliver these interventions. As a result, most LBP care provided in Alberta is "low-value".

With input from Alberta patients, healthcare providers, administrators and international scientists, the Alberta Back Carepathway (ABCp) was designed to overcome these barriers by giving family physicians a common, guideline-based approach to coordinate, assess and manage LBP patients in day-to-day practice.

The ABCp trains family physicians to quickly and easily place patients into 5 categories each having evidence-based interventions that can be provided by physicians at no or low cost to patients and no net cost to the healthcare system. By designing the ABCp to resolve barriers related to training, access and delivery, the ABCp will "pull" rather than "prod" patients and clinicians toward sustained, long-term implementation of this cost-effective solution.

This study is based on a multi-clinic, controlled, non-randomized stepped-wedge study designed for urban and rural primary care networks (PCNs). The primary outcome will be decreased healthcare resource utilization with secondary improvements in quality of life and opioid consumption. Overall, the savings realized through ABCp will create a self-sustaining, scalable solution for LBP care in Alberta.

DETAILED DESCRIPTION:
Justification:

Low back pain (LBP) is a global problem creating more disability than cardiovascular disease and cancer.

In Canada, many people with LBP seek care from general practitioners (GPs) whose services are fully funded by public health programs. Although "free" to Canadians, most approaches used by physicians to address LBP are of low-value - they are often ineffective and potentially dangerous. While research shows that effective LBP interventions are currently available including education, therapeutic exercise, reassurance, manual therapy and non-opioid medications, most LBP patients don't receive these more effective approaches because of their cost (they are not fully funded by public health care) and their GPs are not trained to deliver them. As a result, most LBP patients receive ineffective care that creates 1) unnecessary pain, ongoing disability and potential painkiller addiction, 2) misuse of limited health resources and 3) systemic de-integration of community clinicians who provide evidence-based care for LBP, but are not funded by the current health care system (e.g. Chiropractors and Physical Therapists). To overcome the increasing provision of low-value care for LBP in Canada, the Alberta Back Care pathway has been created (ABCp). The ABCp incorporates GLA:D Back programming (Good Life with Osteoarthritis: Denmark) the elements of which include patient education, structured exercise and data collection. This new program provides evidence-based care at no cost to the patient through innovative decision-making tools that de-medicalize LBP care.

Objectives:

The primary objective is to evaluate the cost-saving performance measures, described by three economic indicators known to be influenced by evidence-based care for LBP. These include 1) the number of LBP visits to family physicians, 2) the number of family physician referrals of LBP patients to specialists and 3) the number of LBP imaging requests from family physicians.

The second objective is to evaluate Quality-Adjusted Life Years (QALY) derived from patient-reported quality of life.

Hypotheses:

the primary outcome will be decreased healthcare resource utilization with secondary improvements in quality of life and opioid consumption. The healthcare resource utilization costs, at both sites, will decrease (a minimal 30% reduction in revisits, imaging and referrals). Overall, the savings realized through ABCp will create a self-sustaining, scalable solution for LBP care in Alberta.

Background:

LBP is a global problem responsible for more years lived with disability than any other condition. As a result, health, societal, and economic burdens associated with LBP approach those of cardiovascular disease, cancer, mental illness, and autoimmune diseases.

While current evidence-based guidelines consistently recommend education, therapeutic exercise and non-opioid medications, these recommendations are infrequently delivered by GPs for many reasons including a lack of incentives and lack of effective implementation strategies. In addition, patients often have preferences for imaging, procedures and referrals and GPs or other clinicians may be complicit in providing ineffective recommendations to appease their patients. Even when first-line treatments are available, they typically require out-of-pocket payment or a health benefit plan thereby severely limiting access for many Canadians. Together, these factors have conspired globally to significantly increase chronic LBP while also increasing use of narcotics, imaging, and specialist referrals.

The ~700,000 annual healthcare visits in Alberta related to LBP illustrate the above problems clearly. Guideline-discordant LBP care accounts for much of the ~$54,000,000 spent on Emergency Departments (ED), Primary Care Networks (PCN) and specialist visits. Guideline-discordant LBP care is not only low value but is potentially harmful. Up to 22% of persons with LBP in Alberta manage their condition with opioids, creating significant risk for opioid use disorder. Potential harms also arise from care delays. Up to 90% of LBP surgical referrals in Alberta never go to surgery which creates consultation wait times of up to 2 years as well as chronicity or additional disability for LBP patients who could benefit from non-invasive interventions. Further, up to 50% of spine imaging is unnecessary which can create nocebo messaging that can initiate or perpetuate care-seeking behavior.

The cost-saving performance measures are described by three economic indicators known to be influenced by evidence-based care for LBP. These include 1) the number of LBP visits to family physicians, 2) the number of family physician referrals of LBP patients to specialists and 3) the number of LBP imaging requests from family physicians.

The second performance measure is Quality-Adjusted Life Years (QALY) derived from patient-reported quality of life using the EQ-5D-5L.

the third performance measure is opioid safety measured by the number of opioid prescriptions dispensed for family physician patients having a diagnosis of LBP. These data will be obtained from the Alberta Pharmaceutical Information Network (PIN) or the College of Physicians and Surgeons of Alberta (CPSA). We will also track dose exposure and duration of use but these will not be tied to costs.

Study design:

A full-scale feasibility trial utilizing a cluster-randomized design in a primary care setting (EWPCN) as well as a secondary care setting (CPC).

METHODS

ABCp methodology Low back pain patients will be assessed by the clinic's physicians using the ABCp. This begins with a 10-minute exam to place LBP patients into Acute, SubAcute, Chronic, Chronic Non-Responsive or Radiculopathy categories.

Each diagnostic category is derived from existing international guidelines and has its own specific prognosis, evidence-based pharmaceutical and non-pharmaceutical interventions and a list of procedures that should be avoided. For patients whose diagnosis category is Sub-Acute, Chronic or stable Radiculopathy, GLA:D Back programs will be funded by the grant at no cost to patients. Overall, two control populations will be used in our design: pre-implementation controls from the 12-months prior to patient enrollment and concurrent controls using clinics who will wait to implement ABCp in Milestone 3.

Overall timeline and setting:

The first 1-6 months (interim stage) will consist of project staging and pre-implementation activities. A project charter consisting of terms of reference for team expectations, accountability and conflict resolution will be completed and ratified by the leadership team and patient advocates. Project infrastructure will be established including approved ethics protocols, operational approvals, REDCap design and testing, creation of a web presence and designing infographics. Following the interim period, clinician training will commence for EWPCN GPs and CPC GLA:D Back clinicians. Training materials will be presented in a form that best suits the team structure and may consist of educational sessions, team seminars, video vignettes, and one-on-one meetings. Frontline staff training will consist of a web-based video that can be accessed at the staff's convenience.

With the completion of pre-implementation activities, full project implementation will begin. The commencement date of enrollment will be flexible to accommodate COVID-19 delays if present. GLA:D Back ban now be provided on a telehealth platform if needed. Enrollment will occur for a period of one year. Once enrollment ends, a one-year follow up period will begin. At completion of enrollment health resource utilization data from the AHS Enterprise Data Warehouse will be obtained for each participant during the 9-month period before they enrolled in the study. Both secondary outcomes (health resource utilization and PROMs) will be compared to traditional concurrent controls (usual care). In total, the duration of the project will be 2.5 years or 30 months (1-6 months pre-implementation activities, 12 months of enrollment, 12 months follow up).

Recruitment:

The EWPCN leadership will identify interested clinics in their jurisdiction and interested clinicians from those clinics will enroll in the study to a maximum of 50% of all clinicians in the PCN.

The CPC leadership will be responsible for enrolling low back pain referrals into ABCp. Those not enrolled will serve as controls.

ELIGIBILITY:
Inclusion Criteria:

* Licensed physicians in the Edmonton West Primary Care Network (EWPCN) and the Calgary Chronic Pain Centre (CPC)
* Age ≥18 years; (no upper age limit)
* English speaking and a resident of Alberta who have cognition and language sufficient to understand written information, and to provide consent.
* Cauda equina syndrome or infection, fracture
* Single or multiple items such as age over 70, female, significant trauma, and prolonged corticosteroid use)
* Cancer (single or multiple items such as older age, and previous history of cancer)
* For the CPC site specifically: additional requirement of depression and anxiety as rated using the PHQ4 exclusion will include score of 3 or greater on the first two questions combined and/or score of 3 or greater on the third and 4th question combined

Exclusion Criteria:

* Low back pain is caused by a recent motor vehicle accident
* WCB case
* Any known contraindication to exercise (i.e., unstable angina, uncontrolled arrhythmia, severe aortic stenosis).
* Current participation in a supervised exercise or rehabilitation program or enrolled in another interventional clinical trial.
* Plans for, or undergoing, surgery that would involve the spine directly or indirectly or place them into a position where any of the interventions in this trial would be contraindicated as a result of the surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-03-31 (Actual); Primary Completion 2027-12-17 (Estimated); Study Completion 2027-12-17 (Estimated)

PRIMARY OUTCOMES:
Primary Care visits | Through study completion, an average of 30 months
  Number of GP revisits for LBP

SECONDARY OUTCOMES:
GP ordered LBP imaging | Through study completion, an average of 30 months
  Diagnostic imaging
GP requested specialist consultations | Through study completion, an average of 30 months
  Number of GP requested specialist consultations

CONTACTS AND LOCATIONS:
Overall Officials: Brandyn Powelske, MScPT, Study Director — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided